CLINICAL TRIAL: NCT05114655
Title: The Effects of Aromatherapy on Stress and Burnout Among Healthcare Providers During the COVID-19 Pandemic: A 3-Arm Randomized, Double Blind, Controlled Trial
Brief Title: Aromatherapy for Stress and Burnout Among Healthcare Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21-10-110
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Stress; Burnout, Professional; Stress, Job
Keywords: aromatherapy; essential oils
MeSH Terms: conditions — Burnout, Professional; Occupational Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 (Experimental): Participants apply an herbaceous, earthy based essential oil blend diluted in fractionated coconut oil to the jawline three times each day for 7 days.
  Interventions: Other: Herbaceous Essential Oil Blend
- Intervention 2 (Experimental): Participants apply a light, citrus-based essential oil blend diluted in fractionated coconut oil to the jawline three times each day for 7 days.
  Interventions: Other: Citrus Essential Oil Blend
- Placebo (Placebo Comparator): Participants apply an inert blend including fractionated coconut oil to the jawline three times each day for 7 days.
  Interventions: Other: Inert Oil

INTERVENTIONS:
Other: Herbaceous Essential Oil Blend — Participants are given a diluted proprietary oil blend of aromatic extracts from resins, bark, and flowers to apply three times daily for the purposes of inhalation.
  Arms: Intervention 1
Other: Citrus Essential Oil Blend — Participants are given a diluted proprietary oil blend of aromatic extracts from citrus peel, and flowers to apply three times daily for the purposes of inhalation.
  Arms: Intervention 2
Other: Inert Oil — Participants are given an inert vegetable based oil blend to apply three times daily for the purposes of inhalation.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential for inhalation of plant-based aromas to reduce stress and burnout among healthcare professionals and staff in hospitals and urgent care centers.

DETAILED DESCRIPTION:
After being informed about the study and potential risks/benefits, participants will provide e-sign informed consent documents and be randomized to one of three groups in a 1:1:1 ratio. Each participant will apply the assigned study oil to the jawline for inhalation three times daily for a total of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-59
* Lives in the United States
* Otherwise healthy
* Employed full time in a capacity that interacts with patients at a hospital, primary, or urgent care center that treats COVID-19 patients. Full time is defined as 35 hours or more each week.

Exclusion Criteria:

* Positive COVID-19 test within 60 days of the study period
* COVID vaccine of any type scheduled during the intervention period or the week prior to the start of the study
* Allergy to any of the ingredients
* Regular smokers in the home (daily or more often)
* Pregnant, trying to conceive, or breastfeeding
* Existing use of an aromatherapy blend for stress management

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Post-intervention score on the Maslach Burnout Inventory for Health Personnel on day 7 | Day 7
  The Maslach Burnout Inventory is a 22-item scale measuring 3 constructs of burnout: emotional exhaustion, depersonalization, and personal achievement. Each item is ranked on a 7-point likert scale, scored from 0-6, with higher scores indicating higher levels of burnout.
Post-intervention score on the Profile of Mood States, abbreviated version on day 7 | Day 7
  The abbreviated version of the profile of mood states contains 40 items across 7 constructs. Each item is scored on a 5 point scale ranging from 0-4 with higher scores indicating higher levels of each construct.
Post-intervention score on the Depression Anxiety Stress Scale (DASS) on day 7 | Day 7
  The DASS is a 42-item scale measuring depression, anxiety, and stress. Each item is measured on a 4-point frequency scale, scored from 0-3, with higher scores indicating greater frequency of each symptom.

CONTACTS AND LOCATIONS:
Locations (1):
- Franklin Health Research Center, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No